CLINICAL TRIAL: NCT04160533
Title: Registry of Arterial Hypertension: "Study of Modern Phenotypes of Arterial Hypertension, Including Secondary Forms, in Order to Create Personalized Methods of Treatment"
Brief Title: Registry of Arterial Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Principal Investigator, Irina E. Chazova, scientific researcher, Department of Hypertension, Institute of Clinical Cardiology named after A.L.Myasnikov, National Medical Research Center of Cardiology of the Ministry of Healthcare of the Russian Federation, Federal State Budgetary Scientific Institution, Research Institute of Cardiology
Other Study IDs: 86
Record Dates: First submitted 2019-08-29; First posted 2019-11-13 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The problem of the quality of primary health care medical system for patients with arterial hypertension is acute for the investigator's country, as these diseases are the most common and cause the high mortality of the population.

The concept of "quality of primary health care medical system" includes its timeliness, accessibility and provision of medical care to the patient at the modern level, which is determined by the degree of performance by doctors of medical and diagnostic measures corresponding current clinical recommendations.

The system of cardiovascular desease registries, established in the Federal State Clinical Hospital of the Russian Federation Ministry of Public Health with the automated analysis of data on examination and treatment, in comparison with clinical Recommendations. It makes possibility to identify shortcomings and develop approaches to improving the provision of medical care to patients in real clinical practice.

Comparative analysis of the quality of examination and treatment in different samples of patients with cardiovascular desease, observed in 2018-2020, compared with results of previous years will identify ptrends in the provision of medical care to patients with cardiovascular desease.

DETAILED DESCRIPTION:
The study will be conducted using the arterial hypertension registry method, which is a computer program with remote access that allows online collection medical data from medical primary care system. To minimize operator errors, doctors was trained before the work with the arterial hypertension registry. User's guide was developed and the rights of users was determined. Data of examination and treatment of patients from 18 years and older with an established diagnosis of hypertension will be added from outpatient cards into the registry of the arterial hypertension. The information is received by the Institution in an impersonal form through a certified dedicated security channel. Patients sign an informed consent for entering their medical data into the registry of arterial hypertension

ELIGIBILITY:
Inclusion Criteria: The diagnosis of arterial hypertension -

Exclusion Criteria: No diagnosis of arterial hypertension

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Study Population: outpatient patients from 18 to 99 years old with a diagnosis of hypertension
Sampling Method: Non-Probability Sample
Enrollment: 10400 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with blood pressure <140/90 mm Hg | 2018 - 2021 years
  The level of systolic and diastolic blood pressure measured according to the rules described in the clinical guidelines for the treatment and diagnosis of arterial hypertension of the European Society of Cardiology during the visit (mmHg) is entered into the database by doctors.

SECONDARY OUTCOMES:
Number of patients with a history of myocardial infarction, chronic renal desease, chronic heart failure, atrial fibrillation. | 2018-2021
  Diagnosis data is entered by doctors as a "yes" or "no" category.
Antihypertensive medications | 2018-2021
  Antihypertensive drugs the patient takes are entered into the database. Drugs are analyzed by groups and daily dosages

CONTACTS AND LOCATIONS:
Locations (17):
- Russia (17):
  - Regional state budgetary institution of health care Altai Regional Cardiology Dispensary State budgetary institution of public health "Volgograd regional clinical hospital No. 1" clinic State budgetary health institution of the Kemerovo region "Kemerovo R, Barnaul, Altayskiy Kray
  - State Healthcare Institution "Engels City Polyclinic No. 2, Engel's
  - State Healthcare Institution "Engels City Polyclinic No. 4, Engel's
  - State budgetary health institution of the Kemerovo region "Kemerovo Regional Clinical Cardiology Dispensary named after Academician L.S. Barbarash, Kemerovo
  - State budgetary institution of the ryazan region "regional clinical cardiological dispensary", Ryazan
  - Municipal budgetary institution of public health "City polyclinic №1" Taganrog Branch №1, Taganrog
  - Municipal budgetary institution of public health "City polyclinic №1" Taganrog Branch №2, Taganrog
  - Municipal budgetary institution of public health "City polyclinic №1" Taganrog Branch №3, Taganrog
  - Municipal budgetary institution of public health "City polyclinic №1" Taganrog Branch №4, Taganrog
  - Municipal budgetary institution of public health "City polyclinic №2" Taganrog Branch №1, Taganrog
  - Municipal budgetary institution of public health "City polyclinic №2" Taganrog Branch №4, Taganrog
  - Municipal budgetary institution of public health services "City ambulance hospital" city of Taganrog, Taganrog
  - State Autonomous Healthcare Institution of the Tyumen Region "Tyumen Institute of Therapy, Tyumen
  - Municipal Health Institution "City Hospital No. 1" Volgodonsk, Volgodonsk
  - Municipal health institution "City polyclinic №1" Volgodonsk, Volgodonsk
  - Municipal health institution "City polyclinic №3" Volgodonsk, Volgodonsk
  - State budgetary institution of public health "Volgograd regional clinical hospital No. 1" clinic, Volgograd